CLINICAL TRIAL: NCT00244738
Title: The Use of Castor Oil as a Labor Initiator in Post-date Pregnancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CASTOR- HMO-CTIL
Record Dates: First submitted 2005-10-26; First posted 2005-10-27 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2005-11

CONDITIONS: Prolonged Pregnancy
Keywords: pregnancy; post-date; induction of labor; castor oil
MeSH Terms: conditions — Pregnancy, Prolonged | interventions — Castor Oil; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Intervention (Active Comparator): Patients who received castor oil for labor induction
  Interventions: Dietary Supplement: Castor oil
- Control (Placebo Comparator): Patients who received sunflower oil as a placebo
  Interventions: Dietary Supplement: Sunflower oil

INTERVENTIONS:
Dietary Supplement: Castor oil — Patients who received castor oil for labor induction
  Arms: Intervention
Dietary Supplement: Sunflower oil — Patients who received sunflower oil as a placebo
  Arms: Control

SUMMARY:
The purpose of the study is to determine whether castor oil is effective in inducing labor.

DETAILED DESCRIPTION:
Castor oil is traditionally given by midwives in order to induce labor. Its efficacy as an initiator of labor was previously tested only in one clinical trial. Unfortunately this study (by Garry et al.) was not sufficiently controlled.

We intent to recruit 84 healthy pregnant women with no contraindication to vaginal delivery that had past their due date. Women will be randomly and blindly divided into equal sized intervention group and control group. Intervention group will be given 60 mL of castor oil in 140 mL of orange juice, while control group will be given a placebo with similar texture. Primary outcome to be tested is the percentage of women entering active labor within 24 hours of administration.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at 40-42 weeks gestation
* Good obstetrical dating
* Singleton
* Intact membranes
* Preinterventional Bishop score less than or equals 4
* No evidence of effective uterine contractions by external tocography
* Living close to hospital

Exclusion Criteria:

* Multiple gestation
* Oligohydramnios or Polyhydramnios
* Abnormal FHR tracing
* Obstetric complication (hypertension, bleeding)
* Ruptured membranes
* Suspected intrauterine growth restriction
* Biophysical score < 8
* Previous cesarean section / myomectomy / Other uterine operation
* Fever, malaise at recruitment
* Chronic illness (renal, hepatic, endocrine)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2006-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Delivery within 24 hours of administering castor oil/placebo | two weeks
  Actual time of delivery

SECONDARY OUTCOMES:
Neonatal apgar scores | 1 minute and 5 minute after delivery
  Neonatal APGAR scores
Umbilical artery pH and Base Excess | Immediately at birth
  Umbilical artery gases
Neonatal complications including hospitalization in NICU | immediately after birth
  Were there any admissions to NICU, what was the reason ?
Mode of delivery (ie. Normal delivery Vs. Cesarean delivery) | Within two weeks of enrollment
  Mode of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Shay Porat, MD, Principal Investigator — Hadassah Medical Organization; Drorit Hochner-Celnikier, MD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Garry D, Figueroa R, Guillaume J, Cucco V. Use of castor oil in pregnancies at term. Altern Ther Health Med. 2000 Jan;6(1):77-9. PMID 10631825